CLINICAL TRIAL: NCT04332887
Title: Effects of a Multidimensional Exercise Program on Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Ai-Fu Chiou, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YM105127F-2
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Surgery; Frailty
Keywords: Cardiac surgery; Frailty; Exercise program; Randomized controlled trial
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Patients in the intervention group will receive a 12-week exercise program including individual nursing consultation, exercise program, nutrition assessment and instructions, and support.
Who Masked: Outcomes Assessor
Masking Description: One research assistant is trained for being a outcomes assessor in this study who did not know the allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multidimensional Exercise Program (Experimental): Patients in the intervention group received a 12-week multidimensional exercise programme that consisted of individual nursing consultation, an exercise program that included moderate intensity walking for 30-45 minutes per day, three days per week and combined resistance exercise, nutrition assessment and instructions, and support.
  Interventions: Behavioral: Multidimensional Exercise Program
- Control group (No Intervention): Patients in this group maintain their daily life activities, and there is no intervention given.

INTERVENTIONS:
Behavioral: Multidimensional Exercise Program — Patients in the experimental group will receive a 12-week multidimensional exercise program; patients in the control group will maintain their usual life activities.
  Arms: Multidimensional Exercise Program

SUMMARY:
This randomized controlled trial study aims to examine the effects of a multidimensional exercise program in cardiac surgery patients. The following hypotheses were tested: patients who received the exercise program will report significant improvement in frailty after the 12-week multidimensional exercise program. Subjects are randomly assigned to the intervention or control group. Patients in the intervention group will receive a 12-week multidimensional exercise program. Data are collected by using medical records and structural questionnaires, measuring handgrip strength, and a four-meter walk test at baseline, 6 weeks, and 12 weeks.

DETAILED DESCRIPTION:
This study aims to develop a multidimensional exercise program and examine the effects of an exercise program on cardiac surgery patients. An experimental design is used. Subjects are recruited using convenience sampling and randomly assigned to the intervention or control group using the block randomization method. Patients in the intervention group will receive a 12-week multidimensional exercise program, including individual nursing consultation, an exercise program that includes moderate intensity walking for 30-45 minutes per day, three days per week combined resistance exercise, nutrition assessment, and instructions, and support. Data are collected by using medical records and structural questionnaires, measuring handgrip strength, and a four-meter walk test at baseline, 6 weeks, and 12 weeks. The data were analyzed using SPSS version 22.0, and data analysis methods include descriptive statistics, independent t-test, chi-square, and generalized estimating equation.

ELIGIBILITY:
Inclusion criteria:

1. aged above 40 years old and received cardiac surgery via median sternotomy with a stable physical condition;
2. at least met one of the frailty phenotypes, including unintentional weight loss, exhaustion, weakness, slow walking speed, and low physical activity proposed by Fried et al. (2001);
3. had clear consciousness (Mini-Mental State Examination score>24) and can communicate with Mandarin or Taiwanese;
4. consent to participate in this study.

Exclusion criteria:

1. bed-ridden, cannot stand or depends on others to complete all activities of daily living;
2. received emergency cardiac surgery;
3. with a mental illness history;
4. had exercise contraindications including: in infectious or acute phases, uncontrolled hypertension, arrhythmia, or diabetes mellitus;
5. had a musculoskeletal disease, which might be aggravated by exercise;
6. participate in phase two of cardiac rehabilitation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-06-02 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Changes in Fried's Phenotype of Frailty Status and Frailty Criteria | baseline, 6week, 12 week
  Changes from baseline Fried's Phenotype of Frailty include five criteria: weight loss, exhaustion, weakness, slowness, and low physical activity at baseline, 6 weeks, and 12 weeks. Each criteria was identified as positive and negative. Frail was defined if more than two criteria were positive. Pre-frail was defined if one criteria was positive.

CONTACTS AND LOCATIONS:
Overall Officials: Ai-Fu Chiou, PhD, Principal Investigator — Professor
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Molino-Lova R, Pasquini G, Vannetti F, Paperini A, Forconi T, Polcaro P, Zipoli R, Cecchi F, Macchi C. Effects of a structured physical activity intervention on measures of physical performance in frail elderly patients after cardiac rehabilitation: a pilot study with 1-year follow-up. Intern Emerg Med. 2013 Oct;8(7):581-9. doi: 10.1007/s11739-011-0654-z. Epub 2011 Jul 9. PMID 21744061
- [Background] Reeves GR, Whellan DJ, O'Connor CM, Duncan P, Eggebeen JD, Morgan TM, Hewston LA, Pastva A, Patel MJ, Kitzman DW. A Novel Rehabilitation Intervention for Older Patients With Acute Decompensated Heart Failure: The REHAB-HF Pilot Study. JACC Heart Fail. 2017 May;5(5):359-366. doi: 10.1016/j.jchf.2016.12.019. Epub 2017 Mar 8. PMID 28285121
- [Background] Waite I, Deshpande R, Baghai M, Massey T, Wendler O, Greenwood S. Home-based preoperative rehabilitation (prehab) to improve physical function and reduce hospital length of stay for frail patients undergoing coronary artery bypass graft and valve surgery. J Cardiothorac Surg. 2017 Oct 26;12(1):91. doi: 10.1186/s13019-017-0655-8. PMID 29073924
- [Background] Gary RA, Cress ME, Higgins MK, Smith AL, Dunbar SB. Combined aerobic and resistance exercise program improves task performance in patients with heart failure. Arch Phys Med Rehabil. 2011 Sep;92(9):1371-81. doi: 10.1016/j.apmr.2011.02.022. PMID 21878207
- [Derived] Huang WT, Liu CY, Shih CC, Chen YS, Chou CL, Lee JT, Chiou AF. Effects of a home-based multicomponent exercise programme on frailty in post-cardiac surgery patients: a randomized controlled trial. Eur J Cardiovasc Nurs. 2025 May 28;24(4):580-592. doi: 10.1093/eurjcn/zvaf014. PMID 39825783